CLINICAL TRIAL: NCT03556891
Title: Pivotal Study of Subcutaneous Tibial Nerve Stimulation With eCoin for Overactive Bladder (OAB) With Urgency Urinary Incontinence (UUI)
Brief Title: Pivotal Study of eCoin for Overactive Bladder With Urgency Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valencia Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111-3281
Record Dates: First submitted 2018-05-22; First posted 2018-06-14 (Actual); Results first posted 2021-07-30 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Overactive Bladder; Urge Incontinence; Incontinence, Urinary; Urinary Urge Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- eCoin Tibial Nerve Stimulation (Experimental)
  Interventions: Device: eCoin Tibial Nerve Stimulation

INTERVENTIONS:
Device: eCoin Tibial Nerve Stimulation — Subcutaneous stimulation of the tibial nerve using the eCoin device.

SUMMARY:
This trial is a prospective, multicenter, single-arm study of the safety and effectiveness of eCoinTM tibial nerve stimulation in subjects having overactive bladder (OAB) with urgency urinary incontinence (UUI). The study will evaluate changes from baseline in OAB symptoms as measured by voiding diaries and patient reported-outcomes through 48 weeks of eCoinTM therapy or 52 weeks of implantation.

DETAILED DESCRIPTION:
This study enrolled and implanted 133 subjects at 15 sites in the US under the original IDE.

Subjects were given the option to extend out to 3 years post activation, with annual visits at 2 and 3 years post activation (96 and 144 weeks post-activation).

Subjects who are still active in the original IDE study will be offered consecutive enrollment in the post approval study and will be given the option to receive a new implant. Subjects who are no longer active, or have exited the study will be given the option to reenter the study and complete two follow-up visits. Subjects re-entering the study will not have the option to receive a new implant. Post approval follow-up of subjects will occur through the year 5 visit (257 weeks post-activation of their original device). Reimplantation of a new eCoin would not reset their follow-up clock.

ELIGIBILITY:
Primary Inclusion Criteria:

1. Women and men between 18 and 80 years old.
2. Diagnosis of overactive bladder with urgency urinary incontinence or mixed urge and stress incontinence with a predominant urgency component (selfreported), for at least 6 months.
3. Individual is without pharmacological treatment of overactive bladder (antimuscarinics and beta-3 agonists).
4. Individual is intolerant of or has an inadequate response to any of anticholinergics, β3-adrenoceptor agonists, onabotulinumtoxinA, or percutaneous tibial nerve stimulation.

Primary Exclusion Criteria:

1. Predominant stress urinary incontinence with more than 1/3 stress urinary incontinent episodes when compared to total urinary incontinent episodes.
2. Clinically significant bladder outlet obstruction.
3. Clinically significant pelvic organ prolapse beyond the hymenal ring.
4. Inadequate skin integrity or any evidence of an infection or inflammation in either lower leg.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-04-12 (Actual); Study Completion 2024-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott MacDiarmid, MD, Principal Investigator — Alliance Urology
Locations (15):
- United States (15):
  - Kaiser Permanente, Downey, California
  - Sequoia Urology Center, Redwood City, California
  - Kaiser Permanente, San Diego, California
  - Sansum Clinic, Santa Barbara, California
  - SurgOne PC, Englewood, Colorado
  - Urology Associates of Norwalk, Norwalk, Connecticut
  - Florida Bladder Institute, Naples, Florida
  - North Shore Medical Group, Skokie, Illinois
  - UnityPoint Clinic, Waterloo, Iowa
  - Chesapeake Urology, Owings Mills, Maryland
  - Adult & Pediatric Urology, Omaha, Nebraska
  - Manhattan Medical Research, New York, New York
  - Alliance Urology Specialists, Greensboro, North Carolina
  - The Institute for Female Pelvic Medicine & Reconstructive Surgery (FPM Institute), Allentown, Pennsylvania
  - South Carolina OB/GYN, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Initial Pivotal Study
Arm/Group | eCoin Tibial Nerve Stimulation
Started | 133
Completed | 120
Not Completed | 13
Not completed — Adverse Event | 4
Not completed — MRI Need | 3
Not completed — Device Failure | 1
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Missing at random | 1
Not completed — Missing due to COVID | 1
Not completed — Protocol Violation | 1
Period: Pivotal Extension Study
Arm/Group | eCoin Tibial Nerve Stimulation
Started | 105
Completed | 41
Not Completed | 64
Period: Pivotal Re-extension
Arm/Group | eCoin Tibial Nerve Stimulation
Started | 31
Completed | 21
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | eCoin Tibial Nerve Stimulation
Number analyzed (Participants) | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 101
  Unknown or Not Reported | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 6
  White | 112
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  United States | 133
Urgency Urinary Incontinence (UUI) Episodes [Mean (Standard Deviation); unit: episodes/day] — Population: Participant with Baseline Urgency Urinary Incontinence (UUI) Episodes of 0 excluded from Intention-to-Treat (ITT) analysis
  episodes/day
    number analyzed (Participants) | 132
    (all) | 4.32 (3.08)
Urinary Voids [Mean (Standard Deviation); unit: voids/day] — Population: Includes patients in the ITT population whose baseline urinary voids value is more than 10 voids per day as prespecified "frequency" group.
  voids/day
    number analyzed (Participants) | 61
    (all) | 13.06 (2.67)
Urgency Episodes [Mean (Standard Deviation); unit: episodes/day] — Population: Participant with Baseline UUI of 0 excluded from ITT analysis
  episodes/day
    number analyzed (Participants) | 132
    (all) | 8.20 (3.65)
Nocturia Episodes [Mean (Standard Deviation); unit: episodes/day] — Population: Participant with Baseline UUI of 0 excluded from ITT analysis
  episodes/day
    number analyzed (Participants) | 132
    (all) | 2.54 (1.04)
Overactive Bladder Questionnaire (OABq) - Short Form [Mean (Standard Deviation); unit: units on a scale] — Range of scale (0-100). Lower is better, thus a decrease from baseline indicates improvement. This is a patient reported outcome questionnaire which asks questions about subjects' symptom severity. Population: 5 participants did not complete OABq at baseline
  units on a scale
    number analyzed (Participants) | 128
    (all) | 66.1 (19.6)
Overactive Bladder Questionnaire (OABq) - Health Related Quality of Life [Mean (Standard Deviation); unit: units on a scale] — Range of scale (0-100). A higher score is better, thus an increase from baseline indicates improvement. This is a patient reported outcome questionnaire in which patients rate various aspects of their quality of life in the context of their condition. Population: 5 participants did not complete OABq at baseline
  units on a scale
    number analyzed (Participants) | 128
    (all) | 45.7 (22.5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Experiencing 50% or Better Improvement in Urgency Urinary Incontinence Episodes as Measured by a 3-day Voiding Diary.
Description: Responder rate
Time Frame: 48 weeks after device activation.
Population: Intent to Treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | eCoin Tibial Nerve Stimulation
Number analyzed (Participants) | 133
percentage of participants | 68 [60 to 76]

2. Primary Outcome: Long-term Safety in All Patients. Percentage of Patients With Device Related Adverse Events.
Description: All adverse events will be reported in all patients up to 52 weeks after implantation.
Time Frame: 52 weeks after implantation.
Population: Intent to Treat plus subject with a baseline UUI of 0.
Measure: Number; unit: percentage of participants
Arm/Group | eCoin Tibial Nerve Stimulation
Number analyzed (Participants) | 133
percentage of participants | 16

3. Secondary Outcome: Moderate-term Safety in All Patients. Percentage of Patients With Device Related Adverse Events.
Description: All adverse events will be reported.
Time Frame: 28 weeks after implantation
Population: Intent to Treat plus subject with a baseline UUI of 0.
Measure: Number; unit: percentage of participants
Arm/Group | eCoin Tibial Nerve Stimulation
Number analyzed (Participants) | 133
percentage of participants | 14

4. Secondary Outcome: Moderate-term Effectiveness Data. Percentage of Subjects Experiencing 50% or Better Improvement in Urgency Urinary Incontinence Episodes as Measured by a 3-day Voiding Diary.
Description: Moderate-term effectiveness data, responder rate
Time Frame: 24 weeks after device activation
Population: Intent to Treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | eCoin Tibial Nerve Stimulation
Number analyzed (Participants) | 133
percentage of participants | 69 [61 to 77]

5. Secondary Outcome: Percentage of Subjects Experiencing 50% or Better Improvement in Urgency Urinary Incontinence Episodes as Measured by a 3-day Voiding Diary
Description: Responder rate
Time Frame: 96 weeks after device activation.
Population: ITT population with available UUI data at 96 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | eCoin Tibial Nerve Stimulation
Number analyzed (Participants) | 69
Percentage of participants | 78 [67 to 87]

6. Secondary Outcome: Percentage of Subjects Experiencing 50% or Better Improvement in Urgency Urinary Incontinence Episodes as Measured by a 3-day Voiding Diary.
Description: Responder rate
Time Frame: 144 weeks after device activation
Population: ITT Population with available UUI data at 144 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | eCoin Tibial Nerve Stimulation
Number analyzed (Participants) | 38
Percentage of participants | 74 [57 to 87]

7. Secondary Outcome: Percentage of Subjects Experiencing 50% or Better Improvement in Urgency Urinary Incontinence Episodes as Measured by a 3-day Voiding Diary.
Description: Responder rate
Time Frame: 205 weeks after device activation
Population: ITT population with available UUI data at 205 weeks.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | eCoin Tibial Nerve Stimulation
Number analyzed (Participants) | 23
Percentage of participants | 61 [39 to 80]

8. Secondary Outcome: Percentage of Subjects Experiencing 50% or Better Improvement in Urgency Urinary Incontinence Episodes as Measured by a 3-day Voiding Diary.
Description: Responder rate
Time Frame: 257 weeks after device activation
Population: ITT population with available UUI data at 257 weeks.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | eCoin Tibial Nerve Stimulation
Number analyzed (Participants) | 21
Percentage of participants | 67 [43 to 85]

9. Secondary Outcome: Long-term Safety in All Patients: Percentage of Patients With Device Related Adverse Events.
Description: All adverse events will be reported in all patients up to 96 weeks after implantation.
Time Frame: 96 weeks after implantation
Population: ITT population
Measure: Number; unit: Percentage of participants
Arm/Group | eCoin Tibial Nerve Stimulation
Number analyzed (Participants) | 133
Percentage of participants | 20

10. Secondary Outcome: Long-term Safety in All Patients: Percentage of Patients With Device Related Adverse Events
Description: All adverse events will be reported in all patients up to 144 weeks after implantation.
Time Frame: 144 weeks after implantation
Population: ITT population
Measure: Number; unit: Percentage of participants
Arm/Group | eCoin Tibial Nerve Stimulation
Number analyzed (Participants) | 133
Percentage of participants | 20

11. Secondary Outcome: Long-term Safety in All Patients. Percentage of Patients With Device Related Adverse Events
Description: All adverse events will be reported in all patients up to 205 weeks after implantation.
Time Frame: 205 weeks after implantation
Population: ITT population
Measure: Number; unit: Percentage of participants
Arm/Group | eCoin Tibial Nerve Stimulation
Number analyzed (Participants) | 133
Percentage of participants | 21

12. Secondary Outcome: Long-term Safety in All Patients. Percentage of Patients With Device Related Adverse Events
Description: All adverse events will be reported in all patients up to 257 weeks after implantation.
Time Frame: 257 weeks after implantation
Population: ITT population
Measure: Number; unit: Percentage of participants
Arm/Group | eCoin Tibial Nerve Stimulation
Number analyzed (Participants) | 133
Percentage of participants | 23

ADVERSE EVENTS:
Time Frame: 257 weeks post-implantation
Description: The analysis set is comprised of "treatment emergent" adverse events, defined as adverse events occurring on or after implantation or attempted implantation of eCoin.
  Importantly, all attempted implantations were successful; thus, the safety results are summarized for all implanted patients.
  At each follow-up visit, patients were asked to report any adverse events and it was recorded on the CRF.
Arm/Group | eCoin Tibial Nerve Stimulation
All-Cause Mortality (participants affected / at risk) | 2/133
Serious Adverse Events (participants affected / at risk) | 4/133
Other Adverse Events (participants affected / at risk) | 40/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | eCoin Tibial Nerve Stimulation (N=133)
Postoperative wound infection (Infections and infestations) | 1 (1)
Implant site infection (Infections and infestations) | 2 (2)
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | eCoin Tibial Nerve Stimulation (N=133)
Device stimulation issue (Product Issues) | 6 (6)
Device dislocation (Product Issues) | 3 (3)
Device malfunction (Product Issues) | 2 (2)
Postoperative wound infection (Infections and infestations) | 7 (7)
Wound abcess (Infections and infestations) | 1 (1)
Incision site erythema (Injury, poisoning and procedural complications) | 2 (2)
Incision site pain (Injury, poisoning and procedural complications) | 5 (5)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 3 (3)
Implant site swelling (General disorders) | 2 (2)
Medical device site discomfort (General disorders) | 1 (1)
Muscoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (2)
Anal incontinence (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
A limitation of the study was the lack of blinding and comparison. Considering that neuromodulation studies are generally not blinded since the therapy itself is sensed, a control group with a similar safety profile to eCoin could not be achieved. We also acknowledge that a 12-month endpoint provides only medium-term data on the durability of response and future longer follow up data will be needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT03556891/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT03556891/SAP_001.pdf